CLINICAL TRIAL: NCT04871646
Title: A Double-blind, Multi-center, Multi-regional, Randomized Controlled, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of CKD-314 in Hospitalized Adult Patients Diagnosed With COVID-19
Brief Title: Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of CKD-314
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A108_02CVD2105
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD-314 (Experimental): Treatment with CKD-314 + SOC
  Interventions: Drug: CKD-314+SOC
- CKD-314 Placebo (Placebo Comparator): Treatment with CKD-314 Placebo + SOC
  Interventions: Drug: CKD-314 Placebo+SOC

INTERVENTIONS:
Drug: CKD-314+SOC — CKD-314 is administered intravenously and standard of care is also performed.
  Arms: CKD-314
Drug: CKD-314 Placebo+SOC — CKD-314 placebo is administered intravenously and standard of care is also performed..
  Arms: CKD-314 Placebo

SUMMARY:
A Double-blind, Multi-center, Multi-regional, Randomized controlled, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of CKD-314 in Hospitalized Adult Patients Diagnosed with COVID-19

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of CKD-314 by comparing the study group and control group in hospitalized adult patients diagnosed with COVID-19 pneumonia

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years
2. Patients diagnosed with COVID-19 infection and pneumonia
3. Patients who have voluntarily decided to participate in the study and signed the informed consent form If a patient cannot provide consent on his or her own, informed consent by a legally authorized representative may be obtained.

Exclusion Criteria:

1. Patients with history of hypersensitivity to the study drug
2. Female patients, either who are or may be pregnant or who are breastfeeding, or female patients of child-bearing potential who are unable to use adequate contraception during the study
3. Patients who are deemed to ineligible to participate in the study for other reasons by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 586 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Time to recovery | From day1 to day 28
  Day of recovery is defined as the first day on which the subject meets the criteria

SECONDARY OUTCOMES:
Time to clinical improvement: Time to clinical improvement (TTCI) | From day1 to day 28
  as time (days) from randomization to a decline of 2 categories on the 8-category ordinal scale of clinical status

CONTACTS AND LOCATIONS:
Overall Officials: Hee Jin Jung, Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No